CLINICAL TRIAL: NCT01716143
Title: Left Atrium Substrate Based Ablation Plus Circumferential Pulmonary Vein Isolation in the Treatment of Persistent and Long-standing Atrial Fibrillation
Brief Title: Left Atrium Substrate Based Ablation Plus Circumferential Pulmonary Vein Isolation to Treat Chronic Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Youquan Wei, Clinical Investigator, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-SR-014
Record Dates: First submitted 2012-10-23; First posted 2012-10-29 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; Mapping
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

ARMS (1):
- catheter ablation (Other)
  Interventions: Procedure: radiofrequency catheter ablation

INTERVENTIONS:
Procedure: radiofrequency catheter ablation

SUMMARY:
The purpose of this study is to determine whether left atrium substrate based ablation plus circumferential is effective in the treatment of persistent and long-standing atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

All persistent or permanent AF patients with refractory or intolerant to at least one Class 1 or Class 3 antiarrhythmic medication.

Exclusion Criteria:

1. Patients with paroxysmal AF (self-terminating episodes lasting < 7 day)
2. Patients who have had a previous AF ablation procedure
3. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The primary study end point was freedom from atrial arrhythmias off antiarrhythmic drugs at 3,6,12,18 and 24 months after a single-ablation. procedure. | 3 years

SECONDARY OUTCOMES:
The percentage of macro-reentrant atrial tachycardia in recurrent arrhythmias after atrial fibrillation ablation | December 31, 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Yang G, Yang B, Wei Y, Zhang F, Ju W, Chen H, Li M, Gu K, Lin Y, Wang B, Cao K, Kojodjojo P, Chen M. Catheter Ablation of Nonparoxysmal Atrial Fibrillation Using Electrophysiologically Guided Substrate Modification During Sinus Rhythm After Pulmonary Vein Isolation. Circ Arrhythm Electrophysiol. 2016 Feb;9(2):e003382. doi: 10.1161/CIRCEP.115.003382. PMID 26857907